CLINICAL TRIAL: NCT01696838
Title: Efficacy of Acupuncture and Moxibustion Treatment in Patients With Quiescent Crohn's Disease:Evaluation With Functional Magnetic Resonance Imaging(fMRI)
Brief Title: Efficacy of Acupuncture and Moxibustion Treatment in Patients With Quiescent Crohn's Disease:Evaluation With fMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHACU-201201
Record Dates: First submitted 2012-09-25; First posted 2012-10-01 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Crohn's Disease; CAM
Keywords: Crohn's disease; acupuncture; moxibustion; fMRI; Gut
MeSH Terms: conditions — Crohn Disease | interventions — Electroacupuncture; Acupuncture Therapy; Moxibustion

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EA group (Experimental): Electroacupuncture group
  Interventions: Other: electroacupuncture; Other: moxibustion
- MOX group (Experimental): Herbs-partitioned moxibustion group
  Interventions: Other: electroacupuncture; Other: moxibustion

INTERVENTIONS:
Other: electroacupuncture — Patients receive electroacupuncture for 30 minutes with a stimulation frequency of 2 /100 Hz and a stimulation intensity varying from 0.1 to 1.0 mA.3 times per week,the duration is 12 weeks.
  Other Names: acupuncture
Other: moxibustion — patients receive herbs-partitioned moxibustion for 2 cones，3 times a week for 12 weeks.
  Other Names: herbs-partitioned moxibustion

SUMMARY:
The purpose of this study is to determine whether acupuncture or moxibustion therapies are effective in the treatment of Crohn's disease. Meanwhile, the investigators aim to evaluate the efficacy by functional magnetic resonance imaging.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether acupuncture or moxibustion therapies are effective in the treatment of Crohn's disease. meanwhile, the investigators aim to evaluate the efficacy by functional magnetic resonance imaging.

Through treating quiescent Crohn's disease by electroacupuncture or moxibustion therapies for 12 weeks, Compare the different brain activation by the different therapies and observe the correlation between brain activation and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50 years;
* right-handed;
* clinical remission (Crohn's Disease Activity Index [CDAI]≤150) for at least 6 months prior to the study;
* C-reactive protein(CRP)<10 mg/l;
* erythrocyte sedimentation rate (ESR) <20 mm/h
* signing awritten informed consent form.

Exclusion Criteria:

* use of corticosteroids and psychotropic medications in the previous 30 days;
* current or prior history of neurological or psychiatric disease based
* on physicians' examination and questionnaires;
* current or prior history of neurosurgery, head injury, cerebrovascular
* insult, or brain trauma involving loss of consciousness;
* learning disability;
* claustrophobia;
* presence of metallic implants in the body;
* being pregnant or during lactation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
CDAI | 1 year
  Crohn's Disease Activity Index

SECONDARY OUTCOMES:
fMRI | 1 year
  Brain activiation tested by BOLD fMRI
IBDQ | 1 year
  Inflammatory Bowel Disease Questionnaire
Inflammatory factors | 1 and a half years
  Intestinal mucosa of IL-6,IL-17,IL-23,etc
Neurotransmitter | 1 and a half years
  5-HT,DA,etc

CONTACTS AND LOCATIONS:
Overall Officials: Wu Huangan, PhD, Study Chair — Shanghai Institute of Acupuncture, Moxibustion and Meridian
Locations (1):
- Shanghai Institute of Acupuncture-Moxibustion and Merdian, Shanghai, Shanghai Municipality, China